CLINICAL TRIAL: NCT05018065
Title: Evaluation of Women's Sexual Functions After Having Covid-19
Brief Title: Sexual Functions and Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma ketenci gencer, Principle investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GaziosmanpasaTREHe
Record Dates: First submitted 2021-08-23; First posted 2021-08-24 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Sexual Behavior
MeSH Terms: conditions — COVID-19; Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 women previously diagnosed with mild - medium Covid-19 and had ambulatory care (Active Comparator): Women sexual dysfunctions were screened using Female Sexual Functioning Index (FSFI)
  Interventions: Behavioral: Women sexual dysfunctions were screened using Female Sexual Functioning Index (FSFI)
- 51 women having no Covid-19 history (Active Comparator): Women sexual dysfunctions were screened using Female Sexual Functioning Index (FSFI)
  Interventions: Behavioral: Women sexual dysfunctions were screened using Female Sexual Functioning Index (FSFI)

INTERVENTIONS:
Behavioral: Women sexual dysfunctions were screened using Female Sexual Functioning Index (FSFI) — sexual dysfunction assesment

SUMMARY:
Sexual health is one the important components of life quality. The aim of this study is to compare sexual dysfunction of women who survived Covid-19 and who didn't undergo Covid-19.

DETAILED DESCRIPTION:
With identifying a new type of coronavirus, the infection disease known as Coronavirus disease-2019 (Covid-19) is still effective worldwide. Within the frame of the description that the health is "a complete physical, mental and social welfare," many physical and mental modality may be expected due to the pandemic and the measures against pandemic. Among them, sexual health is one of the basic indicative factors of human welfare. There are few data on sexual dysfunctions from the previous clinic pandemic experiences. From the very early stages of Covid-19 pandemic, health systems and researches focused on mortalities and short-term morbidities. Although there are similar studies about effects of pandemic on sexual behaviors of general community, there is no comparative study about the effects on sexual functions of women survived from Covid-19 and women having no Covid-19 history, yet. This study aims to compare women survived from Covid-19 and women having no Covid-19 history and having similar characteristics in terms of sexual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed for mild - medium Covid-19 infection and had ambulatory care
* being sexually active

Exclusion Criteria:

* having psychiatric disease
* having any malignity
* having endometriosis
* having a gynecologic surgery history
* having a previous sexual dysfunction

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Sexual function assesment of women previously diagnosed with mild - medium Covid-19 and comparision of results with helath women | 6 months
  Sexual function assesment of women is done by using Female Sexual Functioning Index (FSFI).

CONTACTS AND LOCATIONS:
Locations (1):
- Saglık Bilimleri University Istanbul Gaziosmanpa Trainig and Research Hospital, Istanbul, Turkey (Türkiye)